CLINICAL TRIAL: NCT05137717
Title: A Phase 3, Open-Label, Single-Arm Study to Assess the Efficacy, Safety, and Pharmacokinetics of Maribavir for the Treatment of Cytomegalovirus (CMV) Infection in Japanese Recipients of a Hematopoietic Stem Cell Transplant (HSCT) or Solid Organ Transplant (SOT)
Brief Title: A Study of Maribavir in Japanese People With Cytomegalovirus (CMV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-3001; jRCT2021210056 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-11-25; First posted 2021-11-30 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Cytomegalovirus (CMV)
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Maribavir (Experimental): Maribavir 400 milligrams (mg), tablets, orally twice a day (BID) for up to 8 weeks.
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Maribavir tablets
  Other Names: SHP620; TAK-620

SUMMARY:
The main aim of the study is to check if maribavir can treat Japanese people with Cytomegalovirus (CMV) infection, and to check side effect from the study treatment and how much maribavir participants can take without getting side effects from it.

Japanese recipients of a hematopoietic stem cell transplant (HSCT) or solid organ transplant (SOT) will take Maribavir tablets two times a day for 8 weeks in this study.

During the study, participants will visit their study clinic 18 times as a maximum.

ELIGIBILITY:
Inclusion Criteria

1. Be Japanese with Japanese nationality, >=16 years of age at the time of consent.
2. Be a recipient of HSCT or SOT that is functioning at the time of Screening.
3. Have a documented CMV infection with a screening value of >455 IU/mL in plasma in 2 consecutive assessments, separated by at least 1 day, as determined by a central specialty laboratory qPCR or comparable quantitative CMV DNA results. Both samples should be taken within 14 days prior to first dose of study treatment with the second sample obtained within 5 days prior to first dose of study treatment at Visit 2/Day 0.
4. Have the current CMV infection after HSCT or SOT, either primary or reactivation, which, in the investigator's opinion, requires treatment and have any of the following.

   1. Asymptomatic participants: The subjects do not have CMV tissue-invasive disease or CMV syndrome (SOT subjects only) at Baseline, as determined by the investigator according to the criteria specified by Ljungman et al., 2017.
   2. Refractory or resistant participants: The participant must have a current CMV infection that is refractory to the most recently administered of the anti-CMV treatment agent(s). Refractory is defined as documented failure to achieve >1 log10 (common logarithm to base 10) decrease in CMV DNA level in plasma after a 14 day or longer treatment period with IV ganciclovir/oral valganciclovir, or IV foscarnet.
5. Have all of the following results as part of screening laboratory assessments (results from either the central laboratory or a local laboratory can be used for qualification):

   1. Absolute neutrophil count >=1,000/mm^3 (1.0 × 10^9/L)
   2. Platelet count >=25,000/mm^3 (25 × 10^9/L)
   3. Hemoglobin >=8 g/dL
   4. Estimated creatinine clearance >=30 mL/minute (estimated glomerular filtration rate by Modification of Diet in Renal Disease)
6. Be able to swallow tablets.
7. Have life expectancy of >=8 weeks.
8. Weigh >=40 kg.

Exclusion Criteria

1. Have central nervous system (CNS) CMV tissue-invasive disease or CMV retinitis as assessed by the investigator at the time of Screening and prior to administration at Visit 2/Day 0.
2. Be receiving valganciclovir, ganciclovir, foscarnet, or letermovir when study treatment is initiated, or anticipated to require 1 of these agents during the 8-week treatment period.

   NOTE: Participants receiving letermovir must discontinue 3 days prior to first dose of study treatment. Ganciclovir, valganciclovir, and foscarnet must be discontinued prior to the first dose of study treatment.
3. Have known hypersensitivity to the active substance or to an excipient of the study treatments.
4. Have severe vomiting, diarrhea, or other severe GI illness within 24 hours prior to the first dose of study treatment that would preclude administration of oral medication.
5. Require mechanical ventilation or vasopressors for hemodynamic support at the time of Baseline.
6. Pregnant or nursing female.
7. Have received any investigational agent (including CMV-specific T-cells) with known anti-CMV activity within 30 days before initiation of the study treatment at any time.
8. Have previously received maribavir.
9. Have serum aspartate aminotransferase (AST) >5 times upper limit of normal (ULN) at Screening, or serum alanine aminotransferase (ALT) >5 times ULN at Screening, or total bilirubin >=3.0* ULN at Screening (except for documented Gilbert's syndrome), as analyzed by local or central laboratory.
10. Have known (previously documented) positive results for HIV. Participants must have a confirmed negative HIV test result within 3 months of study entry or, if unavailable, be tested by a local laboratory during the screening period.
11. Have active malignancy with the exception of nonmelanoma skin cancer, as determined by the investigator. Participants who experience relapse or progression of their underlying malignancy (for which HSCT or SOT was performed), as determined by the investigator, are not to be enrolled.
12. Be undergoing treatment for acute or chronic hepatitis C.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- Japan (20):
  - Ehime University Hospital, Tōon, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Imamura General Hospital, Kagoshima, Kagoshima-ken
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Yochomachi Clinic, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Fukushima Medical University Hospital, Fukushima
  - Kyoto University Hospital, Kyoto
  - Okayama University Hospital, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Jichi Medical University Saitama Medical Center, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61a671acf571d4002a64b438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 sites in Japan from 18 January 2022 to 27 June 2023.
Pre-assignment Details: Japanese participants with cytomegalovirus (CMV) infection were enrolled to receive maribavir treatment in this study.
Groups:
- Maribavir: Participants received maribavir 400 milligrams (mg), oral tablet, twice a day (BID) for up to 8 weeks.
Period: Overall Study
Arm/Group | Maribavir
Started | 41
Completed | 33
Not Completed | 8
Not completed — Death | 2
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included of all participants who had taken at least 1 dose of study treatment.
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 41
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 41
Height [Mean (Standard Deviation); unit: centimetres (cm)] | 164.46 (8.702)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 57.47 (10.707)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI was calculated as weight (kg)/ (height [meter]) ^2.
  kilograms per meter square (kg/m^2) | 21.26 (3.538)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Confirmed Clearance of Plasma CMV Deoxyribose Nucleic Acid (DNA) at Week 8
Description: The confirmed viremia clearance was defined as a plasma CMV DNA concentration below the lower limit of quantification (LLOQ) (that is [i.e.], less than [<] 34.5 international units per milliliter [IU/mL]) when assessed by the COBAS® 8800/COBAS® CMV Test, in two consecutive post-baseline samples, separated by at least 5 days. To be considered a responder for the primary endpoint, the participant must have received exclusively study-assigned treatment (regardless of whether study-assigned treatment was completed).
Time Frame: At Week 8
Population: FAS included of all participants who had taken at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maribavir: Participants received maribavir 400 mg, oral tablet, BID for up to 8 weeks.
Arm/Group | Maribavir
Number analyzed (Participants) | 41
percentage of participants | 68.3 [51.9 to 81.9]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: A TEAEs was defined as any event emerging or manifesting at or after the initiation of treatment with an investigational product or medicinal product or any existing event that worsened in either intensity or frequency following exposure to the investigational product or medicinal product. An SAE was any untoward medical occurrence or effect that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability / incapacity, was a congenital anomaly / birth defect or was medically important due to other reasons than the above mentioned criteria.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants
  Participants with TEAEs | 39
  Participants with Serious TEAEs | 13

3. Primary Outcome: Number of Participants With TEAEs Leading to Treatment Discontinuation With Maribavir
Description: The number of participants with TEAEs leading to maribavir study treatment discontinuation (including treatment interruption or withdrawal) were reported.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants | 9

4. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs
Description: Vital sign assessments included blood pressure, pulse, respiratory rate and body temperature. Any clinically meaningful change in vital signs which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Meaningful Abnormalities in Physical Examination Findings
Description: Physical examination included assessments of the head, eyes, ears, nose, throat, neck, lymph nodes, and the cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, genitourinary, and neurological systems. Any clinically meaningful change in physical examination which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Meaningful Abnormalities in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included evaluations of hematology, chemistry, urinalysis. Any clinically meaningful change in clinical laboratory parameters which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Electrocardiograms (ECGs)
Description: 12-lead ECG were evaluated. Any change in ECG assessments which are deemed clinically meaningful by the investigator were reported.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants | 0

8. Primary Outcome: Number of Participants With Events of Immunosuppressant Drug Level Increased in Blood
Description: Immunosuppressant drug concentration testing was solely for participants who received immunosuppressive therapy with tacrolimus, cyclosporine, or everolimus. The number of participants with an increased level of at least one immunosuppressant drug was reported.
Time Frame: From first dose of study drug up to Week 8
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants | 1

9. Primary Outcome: Number of Participants With TEAEs of New Onset of Acute or Chronic Graft-versus-host Disease (GVHD), Graft Rejection, or Graft Loss
Description: New onset of acute or chronic GVHD assessed as TEAEs, and graft rejection, or graft loss assessed were reported.
Time Frame: From first dose of study drug up to Week 20
Population: Safety set included of all participants who had taken at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
Participants
  TEAEs of Acute or Chronic GVHD | 2
  TEAEs of Graft Rejection, or Graft Loss | 0

10. Secondary Outcome: Percentage of Participants Who Maintained CMV Viremia Clearance and CMV Infection Symptom Control at Week 8 Through Weeks 12, 16 and 20
Description: The confirmed viremia clearance was defined as a plasma CMV DNA concentration below the LLOQ (i.e., <34.5 IU/mL) when assessed by the COBAS® 8800/COBAS® CMV Test, in two consecutive post-baseline samples, separated by at least 5 days. Percentage of participants who maintained combined CMV viremia clearance and CMV infection symptom control at Week 8 Through Weeks 12, 16 and 20 were reported.
Time Frame: At Week 8 through Weeks 12, 16 and 20
Population: FAS included of all participants who had taken at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
percentage of participants
  At Week 8 | 68.3 [51.9 to 81.9]
  At Week 12 | 34.1 [20.1 to 50.6]
  At Week 16 | 29.3 [16.1 to 45.5]
  At Week 20 | 26.8 [14.2 to 42.9]

11. Secondary Outcome: Time to First Confirmed CMV Viremia Clearance
Description: Time to first confirmed viremia clearance was defined as time from the start date of first dose of study treatment to the date of confirmed viremia clearance (event), or the date of last CMV DNA assessment on study before the initiation of alternative anti-CMV treatment (censored). The time to first confirmed CMV viremia clearance was calculated as date of first confirmed CMV viremia clearance - randomization date + 1). The date of first confirmed CMV viremia clearance was the date of first of two consecutive samples with plasma CMV DNA <LLOQ that meet the criteria of confirmed CMV viremia clearance.
Time Frame: From first dose of study drug up to Week 20
Population: FAS included of all participants who had taken at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Maribavir
Number analyzed (Participants) | 41
days | 22.0 [15.0 to 23.0]

12. Secondary Outcome: Percentage of Participants With Recurrence of Confirmed CMV Viremia During Follow-up Period in Participants With Confirmed Viremia Clearance at Week 8 Who Required Additional Anti-CMV Treatment
Description: Recurrence of confirmed CMV viremia was defined as plasma CMV DNA concentration greater than or equal to (>= 34.5 IU/mL) LLOQ when assessed by the COBAS® 8800/COBAS®CMV Test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance.
Time Frame: From Week 9 up to Week 20
Population: FAS included of all participants who had taken at least 1 dose of study treatment. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Maribavir
Number analyzed (Participants) | 28
percentage of participants | 42.9

13. Secondary Outcome: Change From Baseline in Plasma CMV Viremia Load
Description: The change from baseline in plasma CMV viral load, i.e., plasma CMV DNA concentration was assessed and reported.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11,12, 14, 16, 18 and 20
Population: FAS included of all participants who had taken at least 1 dose of study treatment. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Maribavir
Number analyzed (Participants) | 38
IU/mL
  Change at Week 1: number analyzed (Participants) | 36
  Change at Week 1 | -0.7821 (0.62350)
  Change at Week 2: number analyzed (Participants) | 35
  Change at Week 2 | -1.4813 (0.71540)
  Change at Week 3: number analyzed (Participants) | 36
  Change at Week 3 | -1.7935 (0.86625)
  Change at Week 4: number analyzed (Participants) | 37
  Change at Week 4 | -1.9555 (0.90538)
  Change at Week 5 | -2.0383 (0.97092)
  Change at Week 6: number analyzed (Participants) | 36
  Change at Week 6 | -1.9922 (1.02593)
  Change at Week 7: number analyzed (Participants) | 33
  Change at Week 7 | -1.9718 (1.10335)
  Change at Week 8: number analyzed (Participants) | 35
  Change at Week 8 | -1.7971 (1.28349)
  Change at Week 9: number analyzed (Participants) | 31
  Change at Week 9 | -1.7771 (0.92825)
  Change at Week 10: number analyzed (Participants) | 30
  Change at Week 10 | -1.6819 (0.93517)
  Change at Week 11: number analyzed (Participants) | 27
  Change at Week 11 | -1.5275 (0.94430)
  Change at Week 12: number analyzed (Participants) | 25
  Change at Week 12 | -1.5383 (1.07532)
  Change at Week 14: number analyzed (Participants) | 20
  Change at Week 14 | -1.7712 (1.08735)
  Change at Week 16: number analyzed (Participants) | 19
  Change at Week 16 | -1.7042 (1.05775)
  Change at Week 18: number analyzed (Participants) | 18
  Change at Week 18 | -1.9569 (0.83577)
  Change at Week 20: number analyzed (Participants) | 18
  Change at Week 20 | -1.9734 (0.91902)

14. Secondary Outcome: Percentage of Participants With Recurrence of CMV Viremia During Study Treatment and in the Follow-Up Period After the Participants Are Discontinued From Study Treatment and While On/Off Study Assigned Treatment
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >= lower limit of quantification (LLOQ, i.e. >=34.5 IU/mL) when assessed by COBAS® 8800/COBAS® CMV Test in 2 consecutive plasma samples at least 5 days apart, after being unquantifiable (<LLOQ, i.e. <34.5 IU/mL) for at least 5 days in 2 consecutive samples during the first 8 weeks of the study. Study Treatment: The first stipulated 8 weeks treatment. Follow up period: period started after completion of stipulated 8 weeks treatment to Week 20. While on study assigned treatment: period over which participants received actual dosing regardless of stipulated 8 weeks completion (Week 8 or earlier). While off study assigned treatment: period after study treatment, regardless of stipulated 8 weeks completion (Week 8 or earlier up to Week 20).
Time Frame: Study treatment: Week 0 to Week 8; Follow-up Period:Week 9 to Week 20; At Any time during study:Week 0 to Week 20; While on study assigned treatment: Week 0 to EOT(Week 8 or earlier); While off study assigned treatment: EOT (Week 8 or earlier) to Week 20
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Maribavir
Number analyzed (Participants) | 36
percentage of participants
  Study Treatment: (Week 0 to Week 8) | 13.9
  Follow-up Period: (Week 9 to Week 20) | 44.4
  At Any Time During the Study (Week 0 to Week 20) | 58.3
  While on Study Assigned Treatment (Week 0 to End of Treatment [EOT] [Week 8 or earlier]) | 8.3
  While off Study Assigned Treatment (EOT [Week 8 or earlier] to Week 20) | 50.0

15. Secondary Outcome: Percentage of Participants With Any Mutations in the CMV Genes Conferring Resistance to Maribavir
Description: Plasma samples were obtained and tested to identify mutations in the viral UL97 and UL54 genes confer resistance to maribavir. Percentage of participants with any mutations in the CMV genes conferring resistance to maribavir was reported.
Time Frame: From first dose of study drug up to Week 20
Population: FAS included of all participants who had taken at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
percentage of participants | 12.2

16. Secondary Outcome: Percentage of Participants Who Achieved Confirmed CMV Viremia Clearance at Week 8 to be Less Than (<) 137 IU/mL
Description: The confirmed CMV viremia clearance at Week 8 was defined as plasma CMV DNA concentrations <137 IU/mL, in 2 consecutive post-baseline samples separated by at least 5 days, regardless of whether study treatment was discontinued before the end of the stipulated 8 weeks of therapy.
Time Frame: At Week 8
Population: FAS included of all participants who had taken at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maribavir
Number analyzed (Participants) | 41
percentage of participants | 73.2 [57.1 to 85.8]

17. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Maribavir
Description: Cmin (pre-dose) of maribavir was assessed.
Time Frame: At Weeks 1, 4, and 8: Pre-dose
Population: Pharmacokinetic set included of all participants in the safety set who had plasma sample drawn and tested for maribavir concentrations. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Maribavir
Number analyzed (Participants) | 36
micrograms per milliliter (mcg/mL)
  Week 1: Pre-dose | 10.08 (105.73)
  Week 4: Pre-dose: number analyzed (Participants) | 31
  Week 4: Pre-dose | 12.31 (108.05)
  Week 8: Pre-dose: number analyzed (Participants) | 29
  Week 8: Pre-dose | 12.37 (95.26)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to Week 20
Description: Safety set included of all participants who had taken at least 1 dose of study treatment.
Arm/Group | Maribavir
All-Cause Mortality (participants affected / at risk) | 2/41
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 26/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maribavir (N=41)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 1
Chronic myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia legionella (Infections and infestations) | 1
Pyrexia (General disorders) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Transplantation complication (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maribavir (N=41)
Anaemia (Blood and lymphatic system disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Generalised oedema (General disorders) | 4
Headache (Nervous system disorders) | 6
Hypertension (Vascular disorders) | 3
Insomnia (Psychiatric disorders) | 4
Nausea (Gastrointestinal disorders) | 10
Neutrophil count decreased (Investigations) | 3
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 6
Taste disorder (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT05137717/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT05137717/SAP_001.pdf